CLINICAL TRIAL: NCT01900431
Title: A Randomized, Double-Masked and Placebo-Controlled Study to Evaluate the Efficacy and Safety of Sarilumab Administered Subcutaneously Every 2 Weeks in Patients With Non-Infectious, Intermediate, Posterior or Pan-Uveitis (NIU)
Brief Title: Phase II Study to Analyze Sarilumab in Non-Infectious Uveitis
Acronym: SARILNIUSATURN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ACT13480; 2012-004845-34; U1111-1130-6500 (Other: UTN)
Record Dates: First submitted 2013-07-11; First posted 2013-07-16 (Estimated); Results first posted 2017-06-20 (Actual); Last update posted 2017-06-20 (Actual); Status verified 2017-05

CONDITIONS: Uveitis
MeSH Terms: conditions — Uveitis | interventions — sarilumab; Prednisone; Methotrexate; Leucovorin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo (for Sarilumab) subcutaneous (SC) injection every 2 weeks (q2w) for 16 weeks during principal treatment period (Part A) with background therapy of Prednisone (or equivalent oral corticosteroid) ≥15 mg/day and <80 mg/day as single therapy or in combination with Methotrexate (MTX) 10 to 25 mg/week and folic acid per local prescribing practice. Responders continued with the same treatment regimen up to Week 50 during extension treatment period (Part B) and non-responders were proposed to be treated with open-label Sarilumab 200 mg q2w in open-label treatment period (Part-C).
  Interventions: Drug: Sarilumab; Drug: Prednisone; Drug: Methotrexate; Drug: Folic/folinic acid; Other: Placebo (for Sarilumab)
- Sarilumab 200 mg q2w (Experimental): Sarilumab 200 mg SC injection q2w for 16 weeks during principal treatment period (Part A) with background therapy of Prednisone (or equivalent oral corticosteroid) ≥15 mg/day and <80 mg/day as single therapy or in combination with MTX 10 to 25 mg/week and folic acid per local prescribing practice. Responders continued with the same treatment regimen up to Week 50 during extension treatment period (Part B) and non-responders were proposed to be treated with open-label Sarilumab 200 mg q2w in open-label treatment period (Part-C).
  Interventions: Drug: Sarilumab; Drug: Prednisone; Drug: Methotrexate; Drug: Folic/folinic acid

INTERVENTIONS:
Drug: Sarilumab — Pharmaceutical form: Prefilled syringes; Route of administration: Subcutaneous
  Other Names: SAR153191/REGN88
Drug: Prednisone — Pharmaceutical form: Tablet or Capsule; Route of administration: Oral
Drug: Methotrexate — Pharmaceutical form: Tablet or Capsule or Suspension; Route of administration: Orally or intravenously or intramuscular
Drug: Folic/folinic acid — Pharmaceutical form: Tablet or Capsule; Route of administration: Oral
Other: Placebo (for Sarilumab) — Pharmaceutical form: Prefilled syringes; Route of administration: Subcutaneous
  Arms: Placebo

SUMMARY:
Primary Objective:

To evaluate the efficacy of sarilumab at Week 16 in participants with non-infectious uveitis (NIU).

Secondary Objectives:

To evaluate the change in best corrected visual acuity (BCVA). To evaluate the safety of subcutaneous sarilumab in participants with NIU. To evaluate the change in macular edema. To evaluate the change in other signs of ocular inflammation. To evaluate the effect on retinal vessel leakage. To evaluate the effect of sarilumab on reducing concomitant immunosuppressant therapy.

To evaluate the change in ocular inflammation in the anterior chamber. To evaluate the pharmacokinetics of sarilumab in NIU participants. To evaluate the immunogenicity with anti-drug antibodies (ADA).

DETAILED DESCRIPTION:
The total duration per participant was up to 58 weeks, which included a 2 week screening period, 16 weeks principal treatment period (Part A), 34 weeks extension treatment period (Part B) or open label treatment period (Part C), and 6 weeks after last treatment administration.

Participants with decrease in vitreous haze (VH) ≥2; or corticosteroids dose <10 mg/day at Week 16 were considered as responders. Participants who did not complete the principal treatment period (Part A) due to lack of efficacy; or no decrease in VH ≥2 and corticosteroids dose ≥10 mg/day at Week 16; or no decrease in VH ≥2 and corticosteroids dose missing at Week 16; or non-responder according to medical review, were considered as non-responders.

Responder participants, observed at Week 16 (at the end of Part A), were invited to continue in the extension treatment period (Part B).

Non-responder participants, observed within the first 16 weeks, were offered to be treated by open-label sarilumab (Part C).

ELIGIBILITY:
Inclusion criteria:

* ≥18 years of age.
* Non-infectious intermediate, posterior, or pan-uveitis in the study eye.
* Active disease at screening or evidence of activity within the 3 months prior to screening visit. Following the approval of amendment-2, only participants with "active disease" as defined above were enrolled in the study.
* Starting oral prednisone dose must be greater than or equal to 15 mg/day and less than 80 mg/day.
* At screening, participants must be receiving oral prednisone (≥15 mg and <80 mg/day [or equivalent oral corticosteroid]) as single immunosuppressive therapy or in combination with MTX (≤25 mg/week) orally or intravenously or intramuscular or subcutaneous). -
* Participants could be receiving one or several of the following therapies: Azathioprine (≤2.5 mg/kg/day), Mycophenolate mofetil (≤2 g daily, orally), Cyclosporine (≤4 mg/kg daily, orally), Tacrolimus (≤4 mg daily, orally).
* The doses might not had been increased for at least 4 weeks prior to the randomization visit.
* At randomization, participants had been receiving oral prednisone (≥15 mg and <80 mg/day [or equivalent oral corticosteroid]) as single immunosuppressive therapy or in combination with MTX (≤25 mg/week) orally or intravenously or intramuscular or subcutaneous).
* Azathioprine, mycophenolate mofetil, cyclosporine and tacrolimus had to be permanently discontinued at least 48 hours prior to the first study treatment injection, or longer as per Investigator's judgment. These immunomodulatory therapies (IMTs) were not permitted anytime during the treatment period.
* Signed written informed consent.

Exclusion criteria:

* Participants with best-corrected visual acuity (BCVA) worse than 20 early treatment diabetic retinopathy study (ETDRS) letters in at least one eye.
* Participants with confirmed or suspected uveitis of infectious etiology or uveitis of traumatic etiology.
* Participants with primary diagnosis of anterior uveitis.
* Prior treatment with anti-interleukin-6 (IL-6) or interleukin-6 receptor complex (IL-6R) antagonist therapies, including tocilizumab and sarilumab.

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2013-10; Primary Completion 2015-07 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (20):
- United States (5):
  - Investigational Site Number 840008, Worcester, Massachusetts
  - Investigational Site Number 840009, Omaha, Nebraska
  - Investigational Site Number 840005, Slingerlands, New York
  - Investigational Site Number 840007, Cleveland, Ohio
  - Investigational Site Number 840006, Arlington, Texas
- Czechia (2):
  - Investigational Site Number 203001, Brno
  - Investigational Site Number 203002, Prague
- France (2):
  - Investigational Site Number 250001, Paris
  - Investigational Site Number 250002, Paris
- Italy (3):
  - Investigational Site Number 380001, Milan
  - Investigational Site Number 380003, Padua
  - Investigational Site Number 380004, Reggio Emilia
- Spain (2):
  - Investigational Site Number 724003, Barcelona
  - Investigational Site Number 724001, Barcelona
- Turkey (Türkiye) (6):
  - Investigational Site Number 792001, Ankara
  - Investigational Site Number 792005, Ankara
  - Investigational Site Number 792002, Istanbul
  - Investigational Site Number 792003, Istanbul
  - Investigational Site Number 792004, Izmir
  - Investigational Site Number 792006, Izmir

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 18 centers in 6 countries. A total of 82 participants were screened between 30 October 2013 and 17 March 2015 of whom 58 participants were randomized and 24 were screen failures. Screen failures were mainly due to exclusion criteria met.
Pre-assignment Details: Participants were randomized in 2:1 ratio (Sarilumab:Placebo) and treated for 16 weeks during principal treatment period (Part A), 30 responders treated up to Week 50 with same dose during extension treatment period (Part B) while 10 non-responders and 11 participants (not completed Part A) treated with open label treatment up to Week 50 (Part C).
Groups:
- Placebo: Placebo (for Sarilumab) subcutaneous (SC) injection every 2 weeks (q2w) for 16 weeks during principal treatment period (Part A) with background therapy of Prednisone (or equivalent oral corticosteroid) ≥15 mg/day and <80 mg/day as single therapy or in combination with Methotrexate (MTX) 10 to 25 mg/week and folic acid per local prescribing practice. Responders continued with the same treatment regimen up to Week 50 during extension treatment period (Part B).
- Sarilumab 200 mg q2w: Sarilumab 200 mg SC injection q2w for 16 weeks during principal treatment period (Part A) with background therapy of Prednisone (or equivalent oral corticosteroid) ≥15 mg/day and <80 mg/day as single therapy or in combination with MTX 10 to 25 mg/week and folic acid per local prescribing practice. Responders continued with the same treatment regimen up to Week 50 during extension treatment period (Part B).
- Sarilumab 200 mg q2w (Open-Label Treatment): Non-responders and non-completers observed in Part A were treated with Sarilumab 200 mg SC injection q2w for 34 weeks as open-label treatment in open-label treatment period (Part C) with background therapy of Prednisone (or equivalent oral corticosteroid) ≥15 mg/day and <80 mg/day as single therapy or in combination with MTX 10 to 25 mg/week and folic acid per local prescribing practice.
Period: Principal Treatment Period (Part A)
Arm/Group | Placebo | Sarilumab 200 mg q2w | Sarilumab 200 mg q2w (Open-Label Treatment)
Started | 20 | 38 | 0
Completed | 13 (8 responders entered Part B and 5 non-responders entered Part C.) | 28 (22 responders entered Part B, 5 non-responders entered Part C, 1 discontinued the study.) | 0
Not Completed | 7 | 10 | 0
Not completed — Adverse Event | 1 | 3 | 0
Not completed — Lack of Efficacy | 6 | 6 | 0
Not completed — Other than specified above | 0 | 1 | 0
Period: Extended Treatment Period (Part B)
Arm/Group | Placebo | Sarilumab 200 mg q2w | Sarilumab 200 mg q2w (Open-Label Treatment)
Started | 8 | 22 | 0
Completed | 7 | 12 | 0
Not Completed | 1 | 10 | 0
Not completed — Adverse Event | 0 | 2 | 0
Not completed — Lack of Efficacy | 1 | 7 | 0
Not completed — Other than specified above | 0 | 1 | 0
Period: Open-Label Treatment Period (Part C)
Arm/Group | Placebo | Sarilumab 200 mg q2w | Sarilumab 200 mg q2w (Open-Label Treatment)
Started | 0 | 0 | 21 (10 non-responders (5 Placebo, 5 Sarilumab) & 11 non-completers (6 Placebo, 5 Sarilumab) from Part A.)
Completed | 0 | 0 | 13
Not Completed | 0 | 0 | 8
Not completed — Adverse Event | 0 | 0 | 2
Not completed — Lack of Efficacy | 0 | 0 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo (for Sarilumab) SC injection q2w for 16 weeks during principal treatment period (Part A) with background therapy of Prednisone (or equivalent oral corticosteroid) ≥15 mg/day and <80 mg/day as single therapy or in combination with MTX 10 to 25 mg/week and folic acid per local prescribing practice. Responders continued with the same treatment regimen up to Week 50 during extension treatment period (Part B) and non-responders were proposed to be treated with open-label Sarilumab 200 mg q2w in open-label treatment period (Part-C).
- Total: Total of all reporting groups
Arm/Group | Placebo | Sarilumab 200 mg q2w | Total
Number analyzed (Participants) | 20 | 38 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.5 (13.0) | 39.3 (15.3) | 40.0 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 23 | 36
  Male | 7 | 15 | 22

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With at Least 2-step Reduction in Vitreous Haze (VH) or Prednisone Dose <10 mg/Day at Week 16
Description: At least 2-step reduction in VH per central review from baseline was evaluated on Miami 9-step scale. VH is the obscuration of fundus by vitreous cells and protein exudation. Each of the 9-step scale (from grade 0 [low opacity] to 8 [more opacity]) images (in increasing order of opacity) are equivalent to approximately 0.3 log units of degradation in visual acuity based on the Bangerter calibration. Participants with prednisone dose <10 mg/day (or equivalent oral corticosteroid) were also evaluated.
Time Frame: Week 16
Population: Modified intent-to-treat population (mITT) included all randomized participants who received at least 1 injection analyzed according to the group to which the participant was allocated by the randomization schedule. Modified multiple imputation approach was used on VH missing adjudicated scores.
Measure: Number; unit: Percentage of participants
Groups:
- Placebo (Part A): Placebo (for Sarilumab) SC injection q2w for 16 weeks during principal treatment period (Part A) with background therapy of Prednisone (or equivalent oral corticosteroid) ≥15 mg/day and <80 mg/day as single therapy or in combination with MTX 10 to 25 mg/week and folic acid per local prescribing practice.
- Sarilumab 200 mg q2w (Part A): Sarilumab 200 mg SC injection q2w for 16 weeks during principal treatment period (Part A) with background therapy of Prednisone (or equivalent oral corticosteroid) ≥15 mg/day and <80 mg/day as single therapy or in combination with MTX 10 to 25 mg/week and folic acid per local prescribing practice.
Arm/Group | Placebo (Part A) | Sarilumab 200 mg q2w (Part A)
Number analyzed (Participants) | 20 | 38
Percentage of participants | 30.0 | 46.1
Statistical Analysis 1: Comparison: Placebo (Part A) vs Sarilumab 200 mg q2w (Part A); Analysis was performed using combined estimate for odds ratio obtained by combining the log-transformation of odds ratio from Cochran Mantel-Haenszel (CMH) analyses of the different imputed datasets, using Rubin's formulae, and then by back-transforming the combined estimate. The CMH analyses were adjusted for randomization stratification factor VH level (VH >= 4 versus VH <4); Test type: Superiority; p = 0.2354, Cochran-Mantel-Haenszel — Threshold for significance at 0.05 level; Odds Ratio (OR) = 2.1, 90% CI 2-sided [0.8 to 5.6] — Sarilumab 200 mg q2w vs Placebo

2. Secondary Outcome: Change From Baseline in VH Scale at Week 16
Description: Change from baseline in VH scale was evaluated on Miami 9-step scale. VH is the obscuration of fundus by vitreous cells and protein exudation. Each of the 9-step scale (from grade 0 [low opacity] to 8 [more opacity]) images (in increasing order of opacity) were equivalent to approximately 0.3 log units of degradation in visual acuity based on the Bangerter calibration. Least squares (LS) mean was calculated using mixed model for repeated measurements (MMRM) model with treatment groups, visits and visit-by-treatment groups interaction as fixed categorical effects as well as fixed continuous covariate of baseline adjudicated VH.
Time Frame: Baseline to Week 16
Population: Analysis was performed on mITT population. Number of participants analyzed = participants with VH assessment at baseline and post-baseline visits.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo (Part A) | Sarilumab 200 mg q2w (Part A)
Number analyzed (Participants) | 13 | 28
units on a scale | -0.1 (0.23) | -0.9 (0.16)
Statistical Analysis 1: Comparison: Placebo (Part A) vs Sarilumab 200 mg q2w (Part A); Analysis was performed using mixed effect model with repeated measures (MMRM) with treatment groups, visits and visit-by-treatment groups interaction as fixed categorical effects, as well as, fixed continuous covariate of baseline adjudicated VH; Test type: Superiority; p = 0.0127, Mixed Models Analysis — Threshold for significance at 0.05 level; Least Square (LS) Mean Difference = -0.7, 90% CI 2-sided [-1.223 to -0.262], Standard Error of Mean 0.29 — Sarilumab 200 mg q2w vs Placebo

3. Secondary Outcome: Percentage of Participants With Anterior Chamber (AC) Cell Score = 0 or At Least 2-step Reduction in Score at Week 16
Description: Participants with AC cell score = 0 or with ≥2 step reduction from baseline at Week 16 were evaluated. Slit lamp examinations were conducted at each visit to assess AC cell count. The number of AC cells observed within a 1 mm × 1 mm slit beam was used to determine the grade according to the Standardization of Uveitis Nomenclature (SUN) criteria: grade 0 = no cells; grade +0.5 = 1 - 5 cells; grade +1 = 6 - 25 cells; grade +2= 26 - 50 cells; grade +3 = too many to count.
Time Frame: Week 16
Population: Analysis was performed on mITT population. Number of participants analyzed = participants with non-missing AC cell score at Week 16.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo (Part A) | Sarilumab 200 mg q2w (Part A)
Number analyzed (Participants) | 15 | 29
Percentage of participants | 86.7 | 86.2
Statistical Analysis 1: Comparison: Placebo (Part A) vs Sarilumab 200 mg q2w (Part A); Analysis was performed using common odds ratio which came from CMH analysis adjusted for randomization stratification factor VH level (VH >=4 versus VH <4); Test type: Superiority; p = 1, Cochran-Mantel-Haenszel — Threshold for significance at 0.05 level; Odds Ratio (OR) = 0.95, 90% CI 2-sided [0.11 to 6.093] — Sarilumab 200 mg q2w vs Placebo

4. Secondary Outcome: Change From Baseline in Best Corrected Visual Acuity (BCVA) Score at Week 16
Description: BCVA score is based on the number of letters read correctly on the Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity chart assessed at a starting distance of 4 meters, and then at 1 meter. The range of ETDRS is 0 to 100 letters. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). An increase in the number of letters read correctly means that vision has improved. LS mean was calculated using MMRM model with treatment groups, randomization strata of VH level (<4, >=4), visits and visit-by-treatment groups interaction as fixed categorical effects, as well as, fixed continuous covariate of baseline BCVA.
Time Frame: Baseline to Week 16
Population: Analysis was performed on mITT population. Number of participants analyzed = participants with BCVA score assessment at baseline and post-baseline visits.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo (Part A) | Sarilumab 200 mg q2w (Part A)
Number analyzed (Participants) | 15 | 29
units on a scale | 3.5 (1.84) | 9.3 (1.36)
Statistical Analysis 1: Comparison: Placebo (Part A) vs Sarilumab 200 mg q2w (Part A); Analysis was performed using MMRM model with treatment groups, randomization strata of VH level (<4, >=4), visits and visit-by-treatment groups interaction as fixed categorical effects, as well as, fixed continuous covariate of baseline BCVA; Test type: Superiority; p = 0.0153, Mixed Models Analysis — Threshold for significance at 0.05 level; LS Mean Difference = 5.8, 90% CI 2-sided [1.99 to 9.67], Standard Error of Mean 2.26 — Sarilumab 200 mg q2w vs Placebo

5. Secondary Outcome: Change From Baseline in Central Retinal Thickness (CRT) At Week 16
Description: CRT was measured by spectral domain optical coherence tomography (SD-OCT), a non-invasive diagnostic system providing high-resolution imaging sections of the retina. All images were transmitted to the central reading center. SD-OCT was performed in the study eye after pupil dilation. LS mean was calculated using MMRM model with treatment groups, randomization strata of VH level (<4, >=4), visits and visit-by-treatment groups interaction as fixed categorical effects, as well as, fixed continuous covariate of baseline CRT.
Time Frame: Baseline to Week 16
Population: Analysis was performed on mITT population. Number of participants analyzed = participants with CRT assessment at baseline and post-baseline visits.
Measure: Least Squares Mean (Standard Error); unit: µm (microns)
Arm/Group | Placebo (Part A) | Sarilumab 200 mg q2w (Part A)
Number analyzed (Participants) | 14 | 29
µm (microns) | -8.9 (11.46) | -35.4 (8.36)
Statistical Analysis 1: Comparison: Placebo (Part A) vs Sarilumab 200 mg q2w (Part A); Analysis was performed using MMRM model with treatment groups, randomization strata of VH level (<4, >=4), visits and visit-by-treatment groups interaction as fixed categorical effects, as well as, fixed continuous covariate of baseline CRT (Automatic measurement from SD-OCT); Test type: Superiority; p = 0.0683, Mixed Models Analysis — Threshold for significance at 0.05 level; LS Mean Difference = -26.5, 90% CI 2-sided [-50.41 to -2.68], Standard Error of Mean 14.2 — Sarilumab 200 mg q2w vs Placebo

6. Secondary Outcome: Percent Change From Baseline in CRT at Week 16
Description: CRT was measured by SD-OCT, a non-invasive diagnostic system providing high-resolution imaging sections of the retina. All images were transmitted to the central reading center. SD-OCT was performed in the study eye after pupil dilation. LS mean was calculated using MMRM model with treatment groups, randomization strata of VH level (<4, >=4), visits and visit-by-treatment groups interaction as fixed categorical effects, as well as, fixed continuous covariate of baseline CRT.
Time Frame: Baseline to Week 16
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo (Part A) | Sarilumab 200 mg q2w (Part A)
Number analyzed (Participants) | 14 | 29
percent change | 0.0 (2.90) | -6.4 (2.15)
Statistical Analysis 1: Comparison: Placebo (Part A) vs Sarilumab 200 mg q2w (Part A); [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.0825, Mixed Models Analysis — Threshold for significance at 0.05 level; LS Mean Difference = -6.4, 90% CI 2-sided [-12.374 to -0.35], Standard Error of Mean 3.55 — Sarilumab 200 mg q2w vs Placebo

7. Secondary Outcome: Percentage of Participants With CRT Thickness <300 Microns at Week 16
Time Frame: Week 16
Population: This endpoint was replaced by the percent change from baseline in CRT at Week 16 as this is more clinically relevant. Zero participant was analyzed.
Arm/Group | Placebo (Part A) | Sarilumab 200 mg q2w (Part A)
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Percentage of Participants Without Retinal Vessel Leakage on Fluorescein Angiography (FA) at Week 16
Time Frame: Week 16
Population: Analysis of this endpoint was not performed as no retinal vessel leakage data was collected at Week 16. Zero participants were analyzed.
Arm/Group | Placebo (Part A) | Sarilumab 200 mg q2w (Part A)
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Percentage of Participants With Prednisone Dose of ≤5 mg/Day (or Equivalent Oral Corticosteroid) at Week 16
Description: Participants with prednisone dose ≤5 mg/day (or equivalent oral corticosteroid) at Week 16 were evaluated.
Time Frame: Week 16
Population: Analysis was performed on mITT population. Number of participants analyzed = participants with non-missing data for prednisone (or equivalent oral corticosteroid) dose at Week 16.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo (Part A) | Sarilumab 200 mg q2w (Part A)
Number analyzed (Participants) | 15 | 29
Percentage of participants | 40.0 | 41.4
Statistical Analysis 1: Comparison: Placebo (Part A) vs Sarilumab 200 mg q2w (Part A); [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 1, Cochran-Mantel-Haenszel — Threshold for significance at 0.05 level; Odds Ratio (OR) = 1.07, 90% CI 2-sided [0.306 to 3.845] — Sarilumab 200 mg q2w vs Placebo

10. Secondary Outcome: Pharmacokinetics (PK) Assessment: Serum Functional Sarilumab Concentration
Description: Serum functional (unbound) sarilumab concentrations were determined using an enzyme-linked immunosorbent assay (ELISA) method with a lower limit of quantification (LLOQ) of 294 ng/mL. Concentrations below LLOQ were set to zero for samples at predose. Post-treatment concentrations below LLOQ were replaced by LLOQ/2. The samples were considered non-eligible for the analysis if the previous dosing time was <11 days or >17 days before the sampling time for every other week regimens.
Time Frame: Predose on Day 1 (Baseline), Week 2, 4, 8, 12, 16, 24, 36, 52, and end of study (EOS) (Week 56)
Population: PK population: all participants who received at least one dose or part of a dose of investigational medicinal product (IMP) with at least one post-dose, non-missing serum concentration value and were analyzed according to treatment actually received. Data of this endpoint was planned to be analyzed for Sarilumab 200 mg q2w arm in Part A and B only.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Sarilumab 200 mg q2w (Part A + Part B): Sarilumab 200 mg SC injection q2w for 16 weeks during principal treatment period (Part A) with background therapy of Prednisone (or equivalent oral corticosteroid) ≥15 mg/day and <80 mg/day as single therapy or in combination with MTX 10 to 25 mg/week and folic acid per local prescribing practice. Responders continued with the same treatment regimen up to Week 50 during extension treatment period (Part B).
Arm/Group | Sarilumab 200 mg q2w (Part A + Part B)
Number analyzed (Participants) | 38
ng/mL
  At Baseline: number analyzed (Participants) | 37
  At Baseline | 0.0 (0.0)
  At Week 2: number analyzed (Participants) | 29
  At Week 2 | 7383.3 (6547.1)
  At Week 4: number analyzed (Participants) | 32
  At Week 4 | 9876.6 (8262.9)
  At Week 8: number analyzed (Participants) | 31
  At Week 8 | 15958.9 (12813.1)
  At Week 12: number analyzed (Participants) | 26
  At Week 12 | 19705.2 (15480.9)
  At Week 16: number analyzed (Participants) | 26
  At Week 16 | 19598.4 (17280.8)
  At Week 24: number analyzed (Participants) | 19
  At Week 24 | 22406.8 (14584.2)
  At Week 36: number analyzed (Participants) | 14
  At Week 36 | 24375.4 (19121.7)
  At Week 52: number analyzed (Participants) | 5
  At Week 52 | 25046.0 (17870.7)
  EOS (Week 56): number analyzed (Participants) | 1
  EOS (Week 56) | 1730.0 (NA) — As only one participant was analyzed at EOS, standard deviation could not be calculated.

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) were collected from signature of the informed consent form up to the final visit (6 weeks after the last treatment administration [Week 56]) regardless of seriousness or relationship to investigational product.
Description: Reported AEs are treatment-emergent adverse events that is AEs that developed/worsened during the 'on treatment period' (time from the first injection of IMP to the last injection of IMP + 6 weeks).
Groups:
- Placebo (Part A + Part B): Placebo (for Sarilumab) SC injection q2w for 16 weeks during principal treatment period (Part A) with background therapy of Prednisone (or equivalent oral corticosteroid) ≥15 mg/day and <80 mg/day as single therapy or in combination with MTX 10 to 25 mg/week and folic acid per local prescribing practice. Responders continued with the same treatment regimen up to Week 50 during extension treatment period (Part B).
- Sarilumab 200 mg q2w (Part A+ Part B): Sarilumab 200 mg SC injection q2w for 16 weeks during principal treatment period (Part A) with background therapy of Prednisone (or equivalent oral corticosteroid) ≥15 mg/day and <80 mg/day as single therapy or in combination with MTX 10 to 25 mg/week and folic acid per local prescribing practice. Responders continued with the same treatment regimen up to Week 50 during extension treatment period (Part B).
- Sarilumab 200 mg q2w: Open-Label Treatment (Part C): Non-responders and non-completers observed in Part A were proposed to be treated with Sarilumab 200 mg SC injection q2w for 34 weeks as open-label treatment in open-label treatment period (Part-C) with background therapy of Prednisone (or equivalent oral corticosteroid) ≥15 mg/day and <80 mg/day as single therapy or in combination with MTX 10 to 25 mg/week and folic acid per local prescribing practice.
Arm/Group | Placebo (Part A + Part B) | Sarilumab 200 mg q2w (Part A+ Part B) | Sarilumab 200 mg q2w: Open-Label Treatment (Part C)
Serious Adverse Events (participants affected / at risk) | 2/20 | 5/38 | 0/21
Other Adverse Events (participants affected / at risk) | 13/20 | 25/38 | 15/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Part A + Part B) (N=20) | Sarilumab 200 mg q2w (Part A+ Part B) (N=38) | Sarilumab 200 mg q2w: Open-Label Treatment (Part C) (N=21)
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Uveitis (Eye disorders) | 0 | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0 | 0
Intraocular pressure increased (Investigations) | 1 | 0 | 0
Liver function test increased (Investigations) | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0
Abortion induced (Surgical and medical procedures) | 0 | 2 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Part A + Part B) (N=20) | Sarilumab 200 mg q2w (Part A+ Part B) (N=38) | Sarilumab 200 mg q2w: Open-Label Treatment (Part C) (N=21)
Neutropenia (Blood and lymphatic system disorders) | 0 | 4 | 1
Cataract (Eye disorders) | 1 | 2 | 0
Retinal infiltrates (Eye disorders) | 1 | 2 | 0
Uveitis (Eye disorders) | 2 | 6 | 1
Visual impairment (Eye disorders) | 1 | 0 | 2
Aphthous ulcer (Gastrointestinal disorders) | 0 | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 3
Nausea (Gastrointestinal disorders) | 1 | 3 | 1
Fatigue (General disorders) | 0 | 3 | 0
Injection site bruising (General disorders) | 0 | 2 | 0
Injection site swelling (General disorders) | 0 | 2 | 0
Pyrexia (General disorders) | 2 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 2 | 0
Bronchitis (Infections and infestations) | 2 | 1 | 0
Ear infection (Infections and infestations) | 0 | 2 | 0
Influenza (Infections and infestations) | 0 | 4 | 2
Nasopharyngitis (Infections and infestations) | 1 | 2 | 6
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 1
Urinary tract infection (Infections and infestations) | 0 | 2 | 2
Accidental overdose (Injury, poisoning and procedural complications) | 4 | 3 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 2 | 1
Alanine aminotransferase increased (Investigations) | 0 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Dizziness (Nervous system disorders) | 0 | 3 | 0
Headache (Nervous system disorders) | 2 | 4 | 2
Hypoaesthesia (Nervous system disorders) | 1 | 2 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 2 | 0
Middle insomnia (Psychiatric disorders) | 0 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Behcet's syndrome (Vascular disorders) | 1 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.